CLINICAL TRIAL: NCT00091338
Title: A Study of Subcutaneous "CYT 99 007" (Interleukin-7) in Conjunction With Peptide Immunization in Patients With Metastatic Melanoma
Brief Title: Interleukin-7 and Vaccine Therapy in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000387802; NCI-04-C-0235; NCT00088322 (obsolete NCT alias)
Record Dates: First submitted 2004-09-07; First posted 2004-09-09 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2005-01

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — MART-1 Antigen; incomplete Freund's adjuvant; Interleukin-7

INTERVENTIONS:
Biological: MART-1 antigen
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant
Biological: recombinant interleukin-7

SUMMARY:
RATIONALE: Interleukin-7 may stimulate a person's white blood cells to kill tumor cells. Vaccines made from peptides may make the body build an immune response to kill tumor cells. Combining interleukin-7 with vaccine therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of interleukin-7 when given with vaccine therapy in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of interleukin-7 (IL-7) when administered with melanoma peptide vaccine emulsified in Montanide ISA-51 in patients with metastatic melanoma.
* Determine the safety of this regimen in these patients.

Secondary

* Determine the biological effects of this regimen on T-cell function and phenotype at various doses and at the optimal biological dose in these patients.
* Determine the pharmacokinetic and pharmacodynamic characteristics of IL-7 in patients treated with this regimen.
* Determine the antitumor effects of IL-7, in terms of a dose-escalation strategy, in these patients.

OUTLINE: This is a dose-escalation study of interleukin-7 (IL-7).

Patients receive IL-7 subcutaneously (SC) on days 0, 3, 6, 9, 12, 15, 18, and 21. Patients also receive melanoma peptide vaccine comprising gp100 antigen and MART-1 antigen emulsified in Montanide ISA-51 SC on days 0, 7, 14, and 21 in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of IL-7 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. After the MTD is determined, an additional 13 patients are treated at that dose level.

Patients are followed at 1, 2, and 5 weeks, at 3 and 6 months, and then at 1 year.

PROJECTED ACCRUAL: A total of 3-37 patients will be accrued for this study within 1-12.3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma

  * Metastatic disease
* Measurable or evaluable disease
* Disease progression during or after prior interleukin-2 (IL-2) OR ineligible to receive high-dose IL-2* OR has disease burden for which IL-2 is not indicated* NOTE: *If patient did not receive prior IL-2, must have progressed after prior standard first-line therapy (e.g., metastasectomy for single lesions or dacarbazine)
* HLA-A*0201-positive disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3*
* Absolute lymphocyte count ≥ 200/mm^3*
* Platelet count > 100,000/mm^3
* No proliferative hematologic disease NOTE: *For 2 consecutive readings performed on 2 different days

Hepatic

* AST and ALT < 3 times upper limit of normal (ULN)
* PT/PTT ≤ 1.5 times ULN
* Hepatitis B negative

  * Positive hepatitis B serology indicative of prior immunization (i.e., positive for antibody against hepatitis B surface antigen AND negative for antibody against hepatitis B core antigen) allowed
* Hepatitis C negative

Renal

* Creatinine ≤ 1.4 mg/dL

Cardiovascular

* Ejection fraction > 45% by MUGA for patients ≥ 50 years of age OR with a history of cardiac disease
* No resting blood pressure > 140/90 mm Hg with standard antihypertensive therapy

Pulmonary

* DLCO/VA and FEV_1 > 50% of predicted on pulmonary function test for smokers OR for patients with clinical evidence of compromised pulmonary function
* No history of severe asthma

Immunologic

* HIV negative
* No history of autoimmune disease
* No splenomegaly

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other medical or psychiatric disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* More than 4 weeks since prior cytokines
* No prior allogeneic hematopoietic stem cell transplantation
* No concurrent growth factors
* No concurrent monoclonal antibodies
* No other concurrent immunotherapy
* No other concurrent cytokines
* No other concurrent biologic agents

Chemotherapy

* See Disease Characteristics
* No prior intensive myeloablative chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* More than 2 weeks since prior systemic corticosteroids for more than 72 hours in duration
* No concurrent systemic steroids

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* No prior splenectomy
* No prior solid organ transplantation

Other

* More than 4 weeks since prior cytotoxic therapy
* No other concurrent cytotoxic therapy
* No concurrent chronic anticoagulation therapy (e.g., high-dose warfarin, heparin, or aspirin)

  * Concurrent low-dose warfarin (1-2 mg) allowed
* No concurrent chronic medication for asthma
* No concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Principal Investigator — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Rosenberg SA, Sportes C, Ahmadzadeh M, Fry TJ, Ngo LT, Schwarz SL, Stetler-Stevenson M, Morton KE, Mavroukakis SA, Morre M, Buffet R, Mackall CL, Gress RE. IL-7 administration to humans leads to expansion of CD8+ and CD4+ cells but a relative decrease of CD4+ T-regulatory cells. J Immunother. 2006 May-Jun;29(3):313-9. doi: 10.1097/01.cji.0000210386.55951.c2. PMID 16699374